CLINICAL TRIAL: NCT07156942
Title: Strategies to Strengthen Physical and Mental Health During Hemodialysis: Rhythm of Life
Brief Title: A Story-Based Game to Reduce Anxiety and Improve Compliance in Hemodialysis Patients: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afra ÇALIK (Other)
Responsible Party: Sponsor-Investigator, Afra ÇALIK, DR, Suleyman Demirel University
Organization: Suleyman Demirel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9566; Scientific Research Projects C (Other: Suleyman Demirel University)
Record Dates: First submitted 2025-05-17; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hemodialysis; Game-Based Learning; Adherence; Anxiety
Keywords: digital game; hemodialysis; adherence; anxiety; serious games
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor (biostatistician) was masked to group assignment. Participants, care providers, and investigators were aware of the assigned interventions. No additional parties were masked in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Story-Based Digital Game (Experimental): Participants in this arm received a short, story-based digital game intervention during their hemodialysis sessions. The game was played once per week for 4 weeks, with each session lasting approximately 10-15 minutes. The game aimed to reduce anxiety, improve treatment adherence, and increase dietary knowledge by engaging patients in interactive scenarios related to dialysis care.
  Interventions: Behavioral: Story-Based Digital Game
- Standard Care (No Intervention): Participants in this arm received standard hemodialysis care without any additional digital game or educational intervention. They followed the usual treatment routines provided by the dialysis unit.

INTERVENTIONS:
Behavioral: Story-Based Digital Game — Participants in this arm played a story-based digital game during their regular hemodialysis sessions. The game was administered once per week, with each session lasting approximately 10 to 15 minutes, over a 4-week period. The game was accessed via an online platform and designed to educate patients on dietary choices, fluid management, and dialysis self-care through interactive storytelling and decision-making tasks.
  Arms: Story-Based Digital Game

SUMMARY:
This clinical study is testing whether a short, story-based digital game played during dialysis can help improve the health and well-being of patients receiving hemodialysis. The researchers believe that using a digital game with an engaging storyline may help reduce anxiety, increase knowledge about healthy eating, and encourage patients to better follow their treatment plans.

The main hypothesis is that this interactive game will lead to lower anxiety levels, better understanding of dietary rules, and higher treatment adherence compared to standard care alone.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 80 years
* Receiving regular hemodialysis treatment for at least 6 months
* Oriented to time, place, and person
* Minimum primary school education
* Able and willing to provide informed consent

Exclusion Criteria:

* Refusal to participate in the study
* Inability to provide informed consent due to cognitive or communication difficulties

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Treatment Adherence Score | Baseline, Week 2, Week 4
  Assessed using the End-Stage Renal Disease Adherence Questionnaire to measure adherence to dialysis schedules and treatment routines.

SECONDARY OUTCOMES:
Change in Dietary Knowledge Score | Baseline, Week 2, Week 4
  Measured using the Hemodialysis Patients' Diet Knowledge Scale.
Change in Anxiety Level | Baseline, Week 2, Week 4
  Assessed using the State Anxiety Inventory (STAI-S) to measure perceived anxiety during treatment.

OTHER OUTCOMES:
Game Experience Score (GAMEX) | Immediately after first game session
  Evaluated only in the intervention group using the Game Experience Questionnaire to assess enjoyment, absorption, and other psychological effects of gameplay.

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study results are currently under consideration for publication, and data sharing may interfere with the peer-review and publication process.

REFERENCES:
- See also: The full version of the game can be accessed online via the link — https://view.genially.com/67b70f2c70b12069df602e8b/interactive-content-basla

DOCUMENTS (3):
  • Study Protocol (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT07156942/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT07156942/SAP_001.pdf
  • Informed Consent Form (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT07156942/ICF_002.pdf